CLINICAL TRIAL: NCT01782794
Title: Measurement of the Changes in Hepatitis B Immunization Coverage in Infants, and the Acceptability Thereof, Before Reimbursement, Then During the Three Years After Reimbursement of InfanrixHexa® in France, Among the General Population
Brief Title: Acceptability of Hepatitis B Vaccination in General Population
Acronym: PopCorn
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113269
Record Dates: First submitted 2013-01-24; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis B
Keywords: Vaccination; Acceptability; General population; Hepatitis B; Vaccine coverage
MeSH Terms: conditions — Hepatitis B | interventions — Data Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: Children aged 12-15 months at the time of the study. Measurements of Hepatitis B vaccination cover prior to InfanrixHexa reimbursement was obtained from this cohort.
  Interventions: Other: Data collection
- Cohort B: Children aged 24-27 months at the time of the study. Measurements of Hepatitis B vaccination cover prior to InfanrixHexa reimbursement was obtained from this cohort.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Poll and questionnaire-based methodology completed by face-to-face interviews, with possible additional follow-up offered to households.

SUMMARY:
The present study is conducted in order to assess the acceptability of Hepatitis B vaccination in French general population before and after reimbursement of the paediatric vaccine InfanrixHexa. Four measurements are planned, first before reimbursement and the others at year 1, 2 and 3 after reimbursement.

DETAILED DESCRIPTION:
The present study aims to evaluate the changes in Hepatitis B immunization coverage and the acceptability thereof among parents, in the general population. This is a national, prospective, epidemiological study, comprising four measurement time-points over a three-year period, (T1 in 2009, T2 in 2010, T3 in 2011, and T4 in 2012) in order to cover the period prior to the introduction of InfanrixHexa® reimbursement, the transition period, and the period following reimbursement of the vaccine. The periods between each data collection time-point will be identical, lasting a year. Two age groups will be investigated at each data collection time-point: 12-15 months and 24-27 months, thus providing measurements before/after reimbursement.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 12 to 15 months or 24 to 27 months inclusive at the time of the study.
* With a parent or legal representative agreeing to take part in the interview.
* Residing in metropolitan France.

Exclusion Criteria:

* Refusal to take part.
* Infants having lived in another country in their first two years of life.

Ages: 12 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of parents (with infants) agreeing to take part in a personal interview.
Sampling Method: Probability Sample
Enrollment: 2413 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Proportion of infants receiving Hepatitis B vaccination. | 4 years

SECONDARY OUTCOMES:
Evaluation of the immunization coverage levels by other vaccines. | 4 years
  The vaccination coverage by other vaccines will be described for each time point (i.e. at the initial time point, and at the years 1, 2 and 3 time points).
Acceptability of vaccinating against Hepatitis B. | 4 Years
  Acceptability of vaccinating against hepatitis B will be evaluated via assessment of the variation of this acceptability amongst parents categorised as "accepting", using their responses to a semi-qualitative questionnaire about vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Gaudelus J, Vie le Sage F, Dufour V, Lert F, Texier N, Pouriel M, Tehard B, Breart G. Public health impact of Infanrix hexa (DTPa-HBV-IPV/Hib) reimbursement: A study programme in France. Part 1: Evolution of hepatitis B vaccine coverage rates in infants aged less than 27 months, in the general population - the PopCorn study. Rev Epidemiol Sante Publique. 2016 Feb;64(1):23-32. doi: 10.1016/j.respe.2015.11.007. Epub 2015 Dec 31. PMID 26748972